CLINICAL TRIAL: NCT03534778
Title: Prognostic Significance of Lymph Node Yield and Lymph Node Ratio in Patients Affected by Squamous Cell Carcinoma of the Oral Cavity, Hypopharynx and Larynx: a Prospective, Multicenter Observational Study
Brief Title: Prognostic Significance of Lymph Node Yield and Lymph Node Ratio Prospective Observational Study
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Roma La Sapienza (Other)
Responsible Party: Principal Investigator, Oreste Iocca, M.D., D.D.S., Researcher, Istituto Clinico Humanitas
Other Study IDs: LNYLNR
Record Dates: First submitted 2018-05-11; First posted 2018-05-23 (Actual); Last update posted 2019-04-19 (Actual); Status verified 2019-04

CONDITIONS: Head and Neck Cancer
MeSH Terms: conditions — Head and Neck Neoplasms | interventions — Lymph Node Ratio

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- patients undergoing neck dissection: all patients undergoing neck dissection
  Interventions: Diagnostic Test: Lymph Node Yield (LNY) and Lymph Node Ratio (LNR)

INTERVENTIONS:
Diagnostic Test: Lymph Node Yield (LNY) and Lymph Node Ratio (LNR) — LNY and LNR will be examined after neck dissection

SUMMARY:
It is still unclear if Lymph Node Yield (LNY) and Lymph Node Ratio (LNR) may have a prognostic role in patients affected by carcinoma of the oral cavity and the oropharynx. Only retrospective studies are available. For this reason, this prospective, multi center, observational study should provide indications in this regard. Proper stratification by patients characteristics will allow to understand if LNY and LNR may enter in the future TNM staging system

DETAILED DESCRIPTION:
Lymph node involvement is a fundamental prognostic factor in head and neck squamous cell carcinoma (SCC). Lymph node yield (LNY), which is the number of lymph nodes retrieved after neck dissection, and lymph node ratio (LNR), which is the ratio of positive lymph nodes out of the total removed, are measurable indicators that may have the potential to be used as prognostic factors. The present study is designed to define the exact role of LNY and LNR regarding the overall and specific survival of patients affected by oral cavity and oropharyngeal SCC.

This is a multicenter study involving tertiary care referral centers in Europe and North America. Patients affected by oral cavity, HPV+ and HPV- oropharyngeal SCC undergoing neck dissection will be consecutively enrolled and followed-up for up to 5 years. Patients and disease characteristic will be properly recorded and centrally analyzed. The primary end-point is to define reliable cut off- values for LNY and LNR which may serve as prognosticators of survival. This will be achieved through the use of ROC curves. Secondary outcomes will be the Overall survival (OS), Disease Specific Survival (DSS), and Progression Free Survival Hazard Ratios (HR) at 2-, 3- and 5 years, which will be evaluated through the Kaplan-Meier method and the difference in survival attested by the log-rank test. Univariate and multivariate analysis will be performed to understand the association of various outcomes with LNY and LNR.

ELIGIBILITY:
Inclusion Criteria:

* patients affected by oral cavity, oropharynx, larynx squamous cell carcinoma

Exclusion Criteria:

* patients affected by other cancers

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients affected by oral or oropharyngeal squamous cell carcinoma who undergo upfront surgery and neck dissection
Sampling Method: Non-Probability Sample
Enrollment: 350 (Estimated)
Dates: Start 2019-01-01 (Actual); Primary Completion 2022-01-01 (Estimated); Study Completion 2024-01-01 (Estimated)

PRIMARY OUTCOMES:
Optimal cut-off value for 5 year Overall Survival | 5 years

CONTACTS AND LOCATIONS:
Locations (1):
- Oreste Iocca, Milan, MI, Italy

REFERENCES:
- [Derived] Iocca O, Farcomeni A, De Virgilio A, Di Maio P, Golusinski P, Malvezzi L, Pellini R, Golusinski W, Rassekh CH, Spriano G. Prognostic significance of lymph node yield and lymph node ratio in patients affected by squamous cell carcinoma of the oral cavity and oropharynx: Study protocol for a prospective, multicenter, observational study. Contemp Clin Trials Commun. 2019 Jan 14;14:100324. doi: 10.1016/j.conctc.2019.100324. eCollection 2019 Jun. PMID 30723839